CLINICAL TRIAL: NCT02769026
Title: Development of Serum, Imaging, and Clinical Biomarker Driven Models to Direct Clinical Management After Pediatric Cardiac Arrest
Brief Title: Prognostication Biomarkers in Pediatric Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ericka Fink, Associate Professor, Pediatric Critical Care Medicine, University of Pittsburgh
Other Study IDs: 1R01NS096714-01A1 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-05-11 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and blood clot stored for future biomarker and DNA analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter study will validate a panel of serum, imaging, and clinical biomarkers to classify patient outcome early after out-of-hospital pediatric cardiac arrest. Results are expected to have a positive and immediate impact in advancing clinical care and outcomes for these children. This work will provide clinicians, families, and researchers with superior tools to assess the severity of brain injury early after resuscitation in order to know who is at risk of brain injury and may benefit from neuroprotective interventions, to monitor response to these interventions, to plan rehabilitation strategy, and to optimize the design of research studies that test novel interventions to improve neurological outcome after cardiac arrest.

DETAILED DESCRIPTION:
Children with cardiac arrest (CA) have mortality rates of 50-90%, largely due to neurological failure as part of the post-resuscitation syndrome. There is a critical gap of knowledge and tools to accurately classify outcome after pediatric CA. Physical examination and laboratory testing inadequately assess the severity of neurologic injury and outcome. Hazards of misclassification include risking adverse effects from ineffective therapies and non-treatment of ostensibly well patients who later are found to have neurologic deficits. Early and accurate identification of the eventual severity of neurologic injury would allow for timely neuroprotective interventions and/or more targeted testing of new therapies in specific risk populations. The long term objective is to improve the neurological outcome of children surviving CA. In this study, investigators will model and validate serum and imaging biomarkers of brain injury with empirical support, and assess their accuracy together with clinical variables in classifying outcome after pediatric CA. The central hypothesis is that serum and imaging biomarkers of brain injury, together with clinical variables, will critically aid in the early classification of favorable outcome after pediatric CA (Vineland Adaptive Behavior Scales score [VABS] > 70) 1 year after pediatric CA in a multicenter prospective study (8-12 centers and 248 subjects). Strong preliminary data supports this hypothesis, and biomarkers will be tested for outcome classification accuracy in the following 3 specific aims:

Aim 1) Serum biomarkers of neuronal (neuron specific enolase and ubiquitin carboxy-terminal hydrolase-L1) and glial injury (S100b and glial fibrillary acidic protein) Aim 2) Regional (occipital-parietal cortex, basal ganglia, and thalamus) brain MRI (T1/T2 and diffusion-weighted imaging) and magnetic resonance spectroscopy (MRS) biomarkers of neuronal injury (N-acetyl-aspartate) and energy failure (lactate) Aim 3 will model the combination of strong serum and imaging biomarkers of brain injury with clinical variables. We will assess serum biomarkers of brain mitochondrial injury with potential for novel therapeutic targets (cardiolipin and oxidized cardiolipin) in an exploratory aim. This proposed research is innovative, because a combined panel of serum and imaging biomarkers with clinical variables to accurately classify outcome after pediatric CA will be prospectively developed and optimized. These proposed aims leverage recent pilot successes and should generate accurate and reliable models of biomarkers that markedly improve post-resuscitation clinical care in children after CA. Furthermore, these results are expected to have a positive impact in advancing neurocritical care for these children, with forthcoming development of a serum biomarker point of care test and biomarker panels that will accurately classify risk of unfavorable outcome for clinicians and researchers needing to stratify by severity of injury, to monitor response to therapy, and ultimately to assist in their rehabilitation and recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 2 weeks -17 years of age
2. Child had an out of hospital CA: defined as "Cessation of cardiac mechanical activity as confirmed by the absence of signs of circulation. Includes the following rhythms: pulseless electrical activity (PEA), asystole, ventricular tachycardia, and ventricular fibrillation" without a specific duration of CA to capture the full breadth of the range of neurological outcomes
3. Children will be admitted to a pediatric or cardiac ICU
4. Children have vascular access for blood draws as part of their standard of care
5. Children have a pre-CA Pediatric Cerebral Performance Category (PCPC) score of 1-3. 6. The caregivers are required to be fluent in English but some sites may support Spanish-speaking only caregivers

Exclusion Criteria:

1. Patients with acute simultaneous brain lesion (trauma, abscess, tumor, bacterial meningitis)
2. Children with do not resuscitate (DNR) status
3. Child is pregnant
4. Child has an absolute or major contraindication for MRI/S (metal in the eyes, cardiac pacemakers, implanted cardioverter defibrillators, neurostimulation systems, and cochlear implants)
5. Child is undergoing brain death evaluation
6. Child has metabolic disease affecting the brain

Ages: 48 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Vineland Adaptive Behavioral Scale [VABS] score | One year from cardiac arrest
  Evaluate serum, imaging, and clinical biomarkers individually and in combined models to classify favorable outcome at 1 year post-CA (Favorable outcome at 1 year post-CA is a VABS score > 70).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fink EL, Clark RSB, Panigrahy A, Berger R, Wisnowski J, Bluml S, Maloney D, Rubin P, Haller T, Bayir H, Beers SR, Kochanek PM, Fabio A; POCCA Investigators. Personalising Outcomes after Child Cardiac Arrest (POCCA): design and recruitment challenges of a multicentre, observational study. BMJ Open. 2020 Oct 27;10(10):e039323. doi: 10.1136/bmjopen-2020-039323. PMID 33109667